CLINICAL TRIAL: NCT07029711
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF RITLECITINIB IN PEDIATRIC PARTICIPANTS 6 TO LESS THAN 12 YEARS OF AGE WITH SEVERE ALOPECIA AREATA
Brief Title: A Study to Learn About Medicine Called Ritlecitinib in Children Aged Between 6 to 12 Years With Severe Alopecia Areata
Acronym: B7981027
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981027; 2024-515438-33-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT05522556 (Available)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Severe Alopecia Areata
Keywords: Alopecia areata; Children; Ritlecitinib
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and their caregivers, Investigators and other site staff will be blinded to their assigned study intervention. Sponsor staff will be blinded to participants' assigned study intervention, except for sponsor staff involved in the assignment or distribution of study intervention and the provision noted below.
  Sponsor staff who are not directly involved with the conduct of this study will prepare analyses and documentation containing unblinded data while the study is ongoing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ritlecitinib higher dose (Experimental): Participants will receive
  1 ritlecitinib higher dose capsule once a day (QD) and 1 placebo lower dose capsule once a day (QD) orally for 24 weeks.
  Interventions: Drug: Ritlecitinib higher dose
- Ritlecitinib lower dose (Experimental): Participants will receive
  1 ritlecitinib lower dose capsule QD and 1 placebo higher dose capsule QD orally for 24 weeks.
  Interventions: Drug: Ritlecitinib lower dose
- Placebo (Placebo Comparator): Participants will receive
  1 placebo higher dose capsule QD and 1 placebo lower dose capsule QD orally for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritlecitinib higher dose — Study intervention will be provided as oral capsules centrally by the sponsor in high-density polyethylene (HDPE) bottles.
  Other Names: Active Treatment
  Arms: Ritlecitinib higher dose
Drug: Ritlecitinib lower dose — Study intervention will be provided as oral capsules centrally by the sponsor in HDPE bottles.
  Other Names: Active Treatment
  Arms: Ritlecitinib lower dose
Drug: Placebo — Study intervention will be provided as oral capsules centrally by the sponsor in HDPE bottles.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called ritlecitinib) for the possible treatment of severe alopecia areata. Alopecia areata is a condition that causes hair loss.

This study is seeking participants who have:

* at least 50% scalp hair loss due to alopecia areata.
* received varicella vaccination (2 doses) or have been infected by varicella zoster virus before based on blood test reports.
* history of clinical response failure to alopecia areata treatment (for children in EU/UK only).

All participants in this study will receive either study medicine (ritlecitinib) or placebo. A placebo does not have any medicine in it but looks just like the medicine being studied.

One-third of participants will receive ritlecitinib higher dose, one-third participants will receive ritlecitinib lower dose, and one-third participants will receive placebo.

The study medicine is a capsule that is taken by mouth. It is taken once each day at home.

The study will compare the experiences of participants receiving ritlecitinib to participants receiving placebo. This will help see if ritlecitinib is safe and effective.

Participants will take part in this study for 6 months. During this time, they will have 8 study visits at the study clinic. The study team will also call participants about 8 times over the phone.

DETAILED DESCRIPTION:
Study B7981027 is being conducted to assess efficacy and safety of ritlecitinib in pediatric participants 6 to <12 years of age with severe AA. The primary objective of this study is to evaluate the efficacy of ritlecitinib compared to placebo in pediatric participants with severe AA on regrowth of lost scalp hair. The secondary objectives are to evaluate safety, tolerability, acceptability and palatability of ritlecitinib and to evaluate the effect of ritlecitinib on patient centered outcomes.

This study will have 3 treatment arms, including 2 ritlecitinib dosage levels (higher and lower doses) and 1 placebo arm. The participants will be assessed for study eligibility at the screening visit after informed consent/assent is obtained (as applicable).

Participants will receive study medication for a duration of 24 weeks.

At least 225 participants will be enrolled in the study. At least 30% of total study population will be recruited from Europe.

The efficacy assessments include Severity of Alopecia Tool (SALT), eyebrow and eyelash assessments. Patient reported outcomes including Patient's Global Impression of Change (PGI-C), Alopecia Areata Patient Priority Outcomes (AAPPO), Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy - Anxiety Short Form 8a and Depressive Symptoms Short Form 6a, Behavior Rating Inventory of Executive Function®, Second Edition (BRIEF®2), and modified Children's Dermatology Life Quality Index (CDLQI) will be assessed throughout the study. Pharmacokinetics of ritlecitinib will be evaluated using sparse sampling.

Safety monitoring will be performed to identify and monitor the known and potential risks of ritlecitinib.

Participants completing the 24-week treatment period of the study may have the option to enter the long-term extension (LTE) Study B7981028, if the eligibility criteria are met. Participants who complete the 24-week treatment period of the study but who are ineligible for the LTE study will undergo a 4-week off-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of AA (including alopecia totalis (AT) and alopecia universalis (AU)) with at least 50% scalp hair loss due to AA (ie, SALT score of ≥50) at both screening and baseline visits, without evidence of terminal hair regrowth within the previous 12 months.
* For study participants in the EU/UK only: History of clinical response failure to AA treatment (such as topical, off-label pharmacologic, or hairpiece prosthetics)
* Documented evidence of having received varicella vaccination (2 doses), OR evidence of prior exposure to varicella zoster virus (VZV) based on serological testing (ie, a positive VZV Immunoglobulin G (IgG) antibody (Ab) result) at screening.

Exclusion Criteria:

* Other (non-AA) types of alopecia, including any known congenital cause of AA.
* Pre-existing hearing loss.
* Any present or history of malignancies or lymphoproliferative disorder such as Epstein-Barr virus (EBV) related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
* Clinically significant depression per PROMIS Parent Proxy Short Form - Depressive symptoms (T-score ≥70).
* Any evidence of untreated or inadequately treated active or latent Mycobacterium tuberculosis (TB) infection; history (one or more episodes) of severe or serious cytomegalovirus (CMV) infection, herpes zoster (shingles) or disseminated herpes simplex; infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Vaccination with live attenuated replication-competent vaccine within 6 weeks of first dose of study intervention.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-05-18 (Estimated)

PRIMARY OUTCOMES:
For US and Countries Following US Analysis Plan: Response based on achieving an absolute Severity of Alopecia Tool (SALT) score ≤20. | Week 24
  The difference in proportions of participants with the SALT ≤20 response at Week 24 between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For EU/UK and Countries Following EU/UK Analysis Plan: Response based on achieving an absolute SALT score ≤10. | Week 24
  The difference in proportions of participants with the SALT ≤10 response at Week 24 between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.

SECONDARY OUTCOMES:
For EU/UK and Countries Following EU/UK Analysis Plan: Patient Global Impression of Change (PGI-C) response defined as a score of "moderately improved" or "greatly improved". | Week 24
  The difference in proportions of participants with the PGI-C response at Week 24 between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Change from baseline (CFB) in SALT score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in means/proportions in the SALT Score at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Response based on achieving absolute SALT score ≤20 at all visits (except for that included as the primary endpoint). | Week 2, Week 4, Week 8, Week 12, Week 18
  The difference in means/proportions in the endpoint at all scheduled time points (except for that included as the primary endpoints) between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Response based on achieving absolute SALT score ≤10 at all visits (except for that included as the primary endpoint). | Week 2, Week 4, Week 8, Week 12, Week 18.
  The difference in means/proportions in the endpoint at all scheduled time points (except for that included as the primary endpoints) between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: PGI-C response at all visits (except for that included as a key secondary endpoint). | Week 2, Week 4, Week 8, Week 12, Week 18.
  The difference in proportions of participants with the PGI-C response at all scheduled time points (except for that included as key secondary endpoint) between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Response based on improvement from baseline for each Alopecia Areata Patient Priority Outcomes (AAPPO) item. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: CFB in Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Depressive Symptoms T-score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: CFB in PROMIS Parent Proxy Anxiety Symptoms T-score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: CFB in BRIEF®2 T-scores for the 3 index scores (Behavior Regulation Index (BRI), Emotion Regulation Index (ERI), Cognitive Regulation Index (CRI)). | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: CFB in modified Children's Dermatology Life Quality Index (CDLQI) total score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Response based on achieving at least 2 grade improvement or a score of 3 in Eyebrow Assessment (EBA) score in participants with an abnormal EBA at baseline. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions of participants with the EBA response at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Response based on achieving at least 2 grade improvement or a score of 3 in Eyelash Assessment (ELA) score in participants with an abnormal ELA at baseline. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions of participants with the ELA response at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Plasma concentration of ritlecitinib. | Post dose hour 1 and hour 3 at day 28 or day 56.
For all countries: Incidence of treatment emergent Adverse Events (AEs). | From the time participant signs informed consent/assent, through and including a minimum of 28 calendar days after the last administration of the study intervention (up to approximately 8 months).
  To evaluate safety and tolerability of ritlecitinib over time.
For all countries: Incidence of Serious Adverse Events (SAEs) and AEs leading to permanent discontinuation from the study. | From the time participant signs informed consent/assent, through and including a minimum of 28 calendar days after the last administration of the study intervention (up to approximately 8 months).
  To evaluate safety and tolerability of ritlecitinib over time.
CFB in AAPPO activity limitation score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.
For all countries: Acceptability and palatability assessment. | Week 2 and Week 18
  To evaluate acceptability and palatability of the age-appropriate formulation.
CFB in AAPPO emotional symptoms score. | Week 2, Week 4, Week 8, Week 12, Week 18, Week 24.
  The difference in proportions/ means in the endpoint at all scheduled time points between each ritlecitinib dose and placebo groups in pediatric AA participants defined by the inclusion and exclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (11):
  - Pediatric Skin Research, Miami, Florida
  - D&H Tamarac Research Center, Tamarac, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Ear, Nose and Throat Consultants, LLC, Omaha, Nebraska
  - Skin Specialists, PC dba Schlessinger MD, Omaha, Nebraska
  - Complete Behavior Health (Dr. Brittany Marshall, Licensed Psychologist), Papillion, Nebraska
  - Northwest Dermatology Institute, Portland, Oregon
  - 3A Research - West Location, El Paso, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - AMR Clinical, Layton, Utah
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China
- Japan (5):
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Kyorin University Hospital, Mitaka, Tokyo
  - Osaka Metropolitan University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
Supporting Information: Study Protocol, SAP, ICF
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981027